CLINICAL TRIAL: NCT00752310
Title: A Phase I, Open-label, Randomized, Crossover Trial in Healthy Subjects Receiving DRV Combined With RTV Low Dose to Compare the Oral Bioavailability of DRV Suspension to That of DRV 300 mg Tablet Under Fasted and Fed Conditions, and to Assess Multiple Dose Pharmacokinetics of the DRV Suspension
Brief Title: TMC114-TiDP29-C169: Bioavailability and Pharmacokinetics Trial Comparing Darunavir Pediatric Suspension Formulation to Current Darunavir Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR012565
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-04

CONDITIONS: Pharmacokinetics
Keywords: TMC114-TiDP29-C169; TMC114-C169; Darunavir (suspension formulation)
MeSH Terms: interventions — Darunavir

INTERVENTIONS:
Drug: Darunavir

SUMMARY:
The purpose of this study is to evaluate in healthy volunteers how much and how fast the new suspension compared to the commercial darunavir tablet, given in combination with low-dose ritonavir, are absorbed into the body (called the relative oral bioavailability).

DETAILED DESCRIPTION:
The objectives of this trial are in Part 1 to compare the rate and extent of absorption of a single oral dose of 600 mg darunavir (DRV) administered as the suspension formulation F051 (under fed and fasted conditions) to that of the commercial tablet formulation F016 (under fed conditions), in the presence of low-dose ritonavir in healthy volunteers; and to compare the rate and extent of absorption of a single oral dose of 600 mg DRV administered as the suspension formulation F051 under fed conditions to that under fasted conditions, in the presence of low-dose ritonavir in healthy volunteers. In Part 2 we want to assess multiple dose pharmacokinetics of DRV administered as the suspension formulation F051 (under fed or fasted conditions, based on the results of Part 1), in the presence of low-dose ritonavir in healthy volunteers. The short-term safety and tolerability of DRV will be evaluated following administration of 3 single oral doses of 600 mg (formulated as suspension and as tablet) and following administration of multiple oral doses (formulated as suspension), all in presence of low-dose ritonavir in healthy volunteers Part 1: during 3 sessions volunteers will orally receive 3 single doses of 600 mg darunavir (DRV): 2 tablets of 300 mg and 6 ml of suspension under fed conditions and 6 mL of suspension (100 mg/mL) under fasted conditions on Day 3. Part 2: subjects will receive DRV suspension, twice daily from Day 1 to 6, with an additional morning dose on Day 7. In Part I rtv 100 mg will be coadministered twice daily from Day 1 to Day 5 and in Part 2 from Day 1 to Day 9.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection
* Normal weight as defined by a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Able to comply with protocol requirements. Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, electrocardiogram (ECG), vital signs, and the results of blood biochemistry, blood coagulation, and hematology tests and a urinalysis carried out at screening.

Exclusion Criteria:

* No positive HIV 1 or HIV 2 test at screening
* no history of significant skin disease such as, but not limited to rash or eruptions, drug allergies, food allergy, dermatitis, eczema, psoriasis, or urticaria
* no history of allergy to drugs such as, but not limited to, sulphonamides and penicillins
* no previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication administered in this trial
* no female subject of childbearing potential without use of effective nonhormonal birth control methods, or not willing to continue practicing these birth control methods for at least 30 days after the end of the treatment period
* no positive pregnancy test or breast feeding at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Part 1: plasma concentrations of DRV and RTV. Time frame day 3: predose and up to 12h, then at 24, 48, 72h. Part 2: plasma concentrations of DRV and RTV. Time frame: predose day 1 and day 5-6; day 7 predose and up to 12h, then at 24, 48, 72h.

SECONDARY OUTCOMES:
Short term safety and tolerability of DRV, formulated as suspension or as tablet, in the presence of low-dose RTV.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: Bioavailability and Pharmacokinetics Trial Comparing Darunavir Pediatric Suspension Formulation to Current Darunavir Tablet — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1004&filename=CR012565_CSR.pdf